CLINICAL TRIAL: NCT07283380
Title: Investigation of the Effect of Two Different Oral Care Methods on Oral Flora and Ventilator Associated Pneumonia in Mechanically Ventilated Patients: A Randomized Controlled Study
Brief Title: Effect of Two Oral Care Methods on Oral Flora and VAP in Mechanically Ventilated Patients
Acronym: ORAVAP-RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AYDIN-VAP-2025-001
Record Dates: First submitted 2025-11-27; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Ventilator Associated Pneumonia ( VAP)
Keywords: Oral Care; Oral Bacterial Colonization; Mechanically Ventilated Patients
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Intervention Model Description: "Patients will be randomly assigned to one of two parallel groups. One group will receive oral care using a pediatric toothbrush, and the other group will receive oral care using a sponge stick. Each patient will receive only the assigned intervention for 5 consecutive days in the intensive care unit. Oral assessments and microbiological samples will be collected to evaluate changes in oral bacterial colonization and the development of ventilator-associated pneumonia (VAP).
Who Masked: Outcomes Assessor
Masking Description: Masking: Single-blind (independent outcome assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pediatric toothbrush group (Experimental): Patients will receive oral care with a pediatric toothbrush for 5 days. Oral swabs and CPIS scores will be monitored.
  Interventions: Device: Pediatric toothbrush
- Sponge stick group (Active Comparator): Patients will receive oral care with a sponge stick for 5 days. Oral swabs and CPIS scores will be monitored.
  Interventions: Device: Sponge stick

INTERVENTIONS:
Device: Pediatric toothbrush — Oral care will be using a pediatric toothbrush for 5 days; oral swabs and CPIS scores will be monitored.
  Arms: Pediatric toothbrush group
Device: Sponge stick — Oral care will be using a sponge stick for 5 days; oral swabs and CPIS scores will be monitored.
  Arms: Sponge stick group

SUMMARY:
This randomized controlled trial aims to evaluate the effect of two oral care methods on oral bacterial colonization and ventilator-associated pneumonia (VAP) in mechanically ventilated intensive care unit (ICU) patients. The study will be conducted in the Anesthesia and General Intensive Care Unit of a hospital in Turkey between October 2025 and June 2026.

A total of 72 patients who meet the inclusion criteria and provide informed consent will be randomly assigned to two groups. Thirty-six patients will receive oral care with a pediatric toothbrush, and 36 patients will receive oral care with a sponge stick, for five consecutive days. Standardized oral care sets containing 0.12% chlorhexidine, recommended for VAP prevention, will be used in both groups.

Oral health and oral care frequency will be assessed daily using the "Oral Care Assessment Scale in Intensive Care Patients (OCAS-ICP)" developed by the researchers. Oral swabs will be collected on Day 1 and Day 6 and analyzed in the microbiology laboratory for colonization with Staphylococcus spp., Pseudomonas spp., and Acinetobacter spp.

The Clinical Pulmonary Infection Score (CPIS) will be used to monitor the development of VAP, including six parameters: fever, leukocytes, tracheal secretions, oxygenation, chest radiography, and culture results. Patients will be evaluated on Days 1 and 6 for changes in oral flora and VAP occurrence.

This study will provide evidence on the effectiveness of different oral care devices in preventing VAP and improving oral health in mechanically ventilated ICU patients.

DETAILED DESCRIPTION:
This study is designed as a randomized controlled trial to evaluate the effect of two different oral care methods on oral bacterial colonization and the incidence of ventilator-associated pneumonia (VAP) in mechanically ventilated patients in the intensive care unit (ICU). The two methods to be compared are oral care performed with a pediatric toothbrush and oral care performed with a sponge stick.

The study population will consist of patients receiving respiratory support with mechanical ventilation in the Anesthesia and General Intensive Care Unit of a hospital in Turkey, between October 2025 and June 2026. A total of 72 patients who meet the inclusion criteria and provide informed consent will be included. Patients will be randomly assigned to one of two groups: 36 patients will receive oral care using a pediatric toothbrush, and 36 patients will receive oral care using a sponge stick, for a period of 5 consecutive days. In both groups, standardized oral care sets containing 0.12% chlorhexidine, a solution recommended for the prevention of VAP, will be used.

Oral assessments and the frequency of oral care are important for effective nursing practices in the ICU. However, there is currently no validated measurement tool in the national or international literature that evaluates both oral and clinical conditions in this patient population. For this reason, the "Oral Care Assessment Scale in Intensive Care Patients (OCAS-ICP)" developed by the researchers, will be applied daily for 5 days to assess the oral health status and oral care needs of patients.

Oral swab samples will be collected from patients on Day 1 (baseline) and Day 6 of the study and evaluated in the microbiology laboratory. The analysis will focus on colonization with bacterial species associated with VAP, specifically Staphylococcus spp., Pseudomonas spp., and Acinetobacter spp. Results will be recorded on the "Microbiology Patient Follow-up Form."

To monitor the development of VAP, the Clinical Pulmonary Infection Score (CPIS) will be used. This scoring system includes six parameters: fever, leukocyte count, tracheal secretions, oxygenation, chest radiograph findings, and culture results. It has been reported that a CPIS score above 6 is highly reliable for diagnosing pneumonia, with 93% sensitivity and 100% specificity. CPIS data will be collected using the "Clinical Pulmonary Infection Score Patient Follow-up Form" within the first 24 hours of ICU admission and during follow-up.

The primary outcomes will be the change in oral bacterial flora and the incidence of VAP between the two study groups. The findings are expected to provide evidence on the effectiveness of different oral care devices in preventing VAP and improving oral health in mechanically ventilated patients in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been on invasive mechanical ventilation for less than 24 hours.
* Patients who provide informed consent through their legal representative or themselves if capable.
* Patients with no prior oral surgery, no head or neck trauma, and no contraindications to oral care.
* Patients aged 18 years or older.

Exclusion Criteria:

* Patients under 18 years of age.
* Patients who have been on mechanical ventilation for more than 24 hours before enrollment.
* Patients with oral surgical procedures or trauma to the head or neck.
* Patients with contraindications to oral care, such as severe oral bleeding, mucositis, or active oral infections.
* Patients or legal representatives who do not provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Mean colony-forming unit (CFU) counts of oral bacterial colonization | Day 1 and Day 6
  Oral swabs are collected from patients on Day 1 and Day 6 and analyzed in the microbiology laboratory to determine the mean CFU counts of Staphylococcus spp., Pseudomonas spp., and Acinetobacter spp. to assess oral bacterial colonization
Incidence of ventilator-associated pneumonia based on the Clinical Pulmonary Infection Score (CPIS) | Day 1 and Day 6
  To monitor the development of ventilator-associated pneumonia, the Clinical Pulmonary Infection Score (CPIS) will be used. This scoring system includes six parameters: body temperature, leukocyte count, tracheal secretions, oxygenation (PaO₂/FiO₂), chest radiograph findings, and microbiological culture results. The total CPIS ranges from 0 to 12, with higher scores indicating worse pulmonary infection and a higher likelihood of ventilator-associated pneumonia. A CPIS score above 6 has been reported to be highly reliable for diagnosing pneumonia, with 93% sensitivity and 100% specificity.

SECONDARY OUTCOMES:
Oral care frequency assessed by the Oral Care Assessment Scale for Intensive Care Patients (OCAS-ICP) | Day 1 to Day 6
  Oral care frequency and oral health status will be assessed using the Oral Care Assessment Scale for Intensive Care Patients (OCAS-ICP). The scale consists of 10 assessment parameters and 17 factors corresponding to these parameters. Each category is scored from 0 to 4 depending on the presence of relevant factors. The total score obtained from the scale ranges from 0 to 26, with higher scores indicating poorer oral health status and a greater presence of risk factors, and lower scores indicating better oral health status. Patients will be evaluated daily during their intensive care unit stay. Based on the total OCAS-ICP score, oral care will be planned and implemented as follows: patients with a total score of 0-8 points will receive oral care twice daily (2×1), those with 9-17 points will receive oral care four times daily (4×1), and those with 18-26 points will receive oral care six times daily (6×1).Patients will be evaluated daily from Day 1 to Day 6.

CONTACTS AND LOCATIONS:
Overall Officials: Gulten OKUROĞLU, Assoc.Prof, Principal Investigator — Marmara University; Ayse AYDIN, PhDCand., Study Director — Marmara University
Locations (2):
- Turkey (Türkiye) (2):
  - Zonguldak Ataturk State Hospital, Zonguldak
  - Zonguldak Atatürk State Hospital, Ministry of Health, Türkiye, Zonguldak

IPD SHARING:
Plan to Share IPD: No
The decision regarding individual participant data (IPD) sharing has not yet been made. Due to ethical considerations and patient confidentiality concerns in critically ill populations, the research team remains undecided about whether de-identified data can be made available in the future.

REFERENCES:
- [Result] Diaconu O, Siriopol I, Polosanu LI, Grigoras I. Endotracheal Tube Biofilm and its Impact on the Pathogenesis of Ventilator-Associated Pneumonia. J Crit Care Med (Targu Mures). 2018 Apr 1;4(2):50-55. doi: 10.2478/jccm-2018-0011. eCollection 2018 Apr. PMID 30581995
- [Result] Miranda AF, de Paula RM, de Castro Piau CG, Costa PP, Bezerra AC. Oral care practices for patients in Intensive Care Units: A pilot survey. Indian J Crit Care Med. 2016 May;20(5):267-73. doi: 10.4103/0972-5229.182203. PMID 27275074
- [Result] Terezakis E, Needleman I, Kumar N, Moles D, Agudo E. The impact of hospitalization on oral health: a systematic review. J Clin Periodontol. 2011 Jul;38(7):628-36. doi: 10.1111/j.1600-051X.2011.01727.x. Epub 2011 Apr 7. PMID 21470276
- See also: Endotracheal Tube Biofilm and its Impact on the Pathogenesis of Ventilator-Associated Pneumonia — https://pubmed.ncbi.nlm.nih.gov/30581995/
- See also: Oral care practices for patients in Intensive Care Units: A pilot survey — https://pubmed.ncbi.nlm.nih.gov/27275074/
- See also: The impact of hospitalization on oral health: a systematic review — https://pubmed.ncbi.nlm.nih.gov/21470276/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT07283380/Prot_SAP_000.pdf
  • Informed Consent Form (2025-09-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT07283380/ICF_001.pdf